CLINICAL TRIAL: NCT00444743
Title: A Phase 2, Double - Blind, Placebo - Controlled, Randomized Study to Evaluate the Tolerability, Pharmacokinetics, Pharmacodynamics, and Biologic Activity of MM-093 in Patients With Moderate to Severe Uveitis
Brief Title: Phase 2 Study of MM-093 to Treat Patients With Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Merrimack Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MM-093-03-200; IND #100,184
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: MM-093
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MM-093 — 60 mg, administered subcutaneously, weekly
  Arms: 1
Other: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the tolerability, pharmacokinetics, pharmacodynamics, and biologic activity of MM-093 in patients with moderate to severe uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol - specific procedures being performed.
* Have been diagnosed with sarcoid or birdshot uveitis
* Be able and willing to comply with study visits and procedures per protocol.
* Women of child bearing potential must use medically acceptable means of birth control in an effective manner and agree to continue its use during the study and 6 weeks after the last dose of study drug.
* Sexually active men must agree to use a medically acceptable form of contraception during the study and continue for 4 weeks after the last dose of study drug.
* Able to store patient kit/cooler containing study drug in a refrigerator at home.

Exclusion Criteria:

* Significant concurrent medical diseases including:

  * Cancer or history of cancer, or lymphoproliferative disorder (other than sarcoidosis or successfully resected cutaneous basal or squamous cell carcinoma) within 5 years before the screening visit.
  * Any condition for which participation in this study is judged by the physician to be detrimental to the patient, such as history of significant or unstable cardiac, pulmonary, gastrointestinal, neurological, or psychiatric disease.
  * Significant ongoing infection requiring systemic antibiotic, antifungal, antiviral, or ant anti-mycobacterial therapy.
* Autoimmune or connective tissue disorder other than sarcoid or birdshot uveitis, (e.g. Rheumatoid Arthritis, Systemic Lupus Erythematosus, or Scleroderma.)
* Other known active eye diseases or eye infections (bacterial, fungal, or viral) that may interfere with the evaluation of uveitis.
* Grade 2 or above liver function abnormality
* Renal disease
* Any previous history of immunodeficiency syndromes or infection with human immunodeficiency virus (HIV), or a history of hepatitis C or chronic hepatitis B.
* Live viral or bacterial vaccinations within 3 months prior to screening, or planning to receive such vaccinations during the trial, or up to 3 months after the last injection of MM-093.
* Pregnant or breastfeeding women or women planning to become pregnant during the study or within 4 weeks after the last dose of the study drug.
* Scheduled elective surgery during study participation
* Participated in any previous clinical trials using MM-093 or have any prior exposure to MM-093.
* History of severe hypersensitivity to goat, sheep, or cow milk products derived from goat, sheep or cow milk (patients who are lactose intolerant are not excluded.)
* Any other acute or clinically important condition that the investigator feels would jeopardize the integrity of the study (e.g. a CTCAE grade 2 or above clinical finding or laboratory result.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MM-093, as compared to placebo, when administered as a monotherapy once a week for 24 weeks after discontinuing IMT therapy.
To evaluate the biological activity of MM-093, as compared to placebo, as defined by the proportion of patients who have a relapse in their uveitis after discontinuing IMT therapy.

SECONDARY OUTCOMES:
To evaluate the time to relapse of uveitis after IMT therapy has been discontinued.
To evaluate the degree of IMT tapering before a recurrence of uveitis occurs.
To evaluate visual function as evidenced by visual acuity and by electroretinography.
To evaluate sub clinical inflammation as measured by fluorescein angiography.
To evaluate the formation of anti-MM-093 antibodies after MM-093 administration.
To evaluate the formation of anti-goat antibodies after MM-093 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Stephen Foster, Principal Investigator — Massachusetts Eye Research and Surgery Institute
Locations (1):
- MERSI, Cambridge, Massachusetts, United States